CLINICAL TRIAL: NCT06214221
Title: A Randomized Controlled Trial Evaluating the Safety and Effectiveness of the Intelligently-Driven Signos System for Personalized Weight Management in Overweight and Obese Adults
Brief Title: Using Signos mHealth Platform in Adults for Weight Management
Acronym: SWEET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Signos Inc (Industry)
Collaborators: Lindus Health, Inc. (Unknown)
Responsible Party: Principal Investigator, Stephanie Kim, M.D., MPH, Clinical Trial Investigator, Signos Inc, Signos Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIGNOS-CGM-SWEET-301-2023
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Overweight and Obesity; Metabolic Syndrome; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Intervention Model Description: In an open-label randomization model, participants and researchers both know the treatment each participant is receiving. This model involves randomly assigning participants to different treatment groups, ensuring unbiased distribution across interventions, but without concealing the nature of the treatment from either the participants or the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Signos System (Experimental): For all consented participants, the Signos app will use CGM data to provide recommendations customized to users for promoting general health and wellness.
  Interventions: Device: Signos System
- Standard Lifestyle Education (Active Comparator): The "Active Comparator: Standard Lifestyle Education" arm in the clinical trial refers to a control group that receives conventional lifestyle modification advice instead of the experimental Signos System.
  Interventions: Other: Standard Lifestyle Education

INTERVENTIONS:
Device: Signos System — The intervention involves the use of the Signos System, a combination of a proprietary software application with a continuous glucose monitor (CGM), to manage weight in overweight and obese adults.
  Arms: Signos System
Other: Standard Lifestyle Education — In the "Standard Lifestyle Education" arm, participants receive conventional advice on diet and exercise, focusing on general healthy lifestyle habits to manage weight.
  Arms: Standard Lifestyle Education

SUMMARY:
Metabolic syndrome and resulting downstream health effects remains a growing health concern. In published trials, the use of continuous glucose monitoring (CGM) assists behavioral changes efforts, leading to improved adherence and results from diet and exercise changes in individuals with obesity. Mobile health (mHealth) platforms provide satisfactory, easy-to-use tools that help participants in the pursuit of weight change goals. The investigators hypothesize that the use of CGM data and targeted coaching and nutrition education will assist with weight optimization goals in the general (non-diabetic) population using the Signos mHealth platform, with associated health benefits.

DETAILED DESCRIPTION:
The scope of this study is to enroll participants into a study that utilizes a continuous glucose monitor (CGM) and mobile health application [Signos] to optimize general wellness and body weight and composition. The Signos users will be compared against a control arm.

ELIGIBILITY:
Inclusion Criteria:

To join our study, participant need to:

* Be at least 22 years old.
* Be overweight or obese, which we define as having a Body Mass Index (BMI) between 25 and 40.
* HbA1c test result should be below 6.5% at the start of the study.
* Have and know how to use a smartphone that's compatible with the Signos app.
* Be able to understand, speak, and read English well enough to participate fully in the study.

Exclusion Criteria:

Participant can't join our study if participant has:

* Have Type 1 or Type 2 diabetes.
* Are already using a device to monitor glucose level.
* Have severe allergies to the sticky part of glucose monitors.
* Suffer from an eating disorder like anorexia or bulimia.
* Are currently taking certain medications for diabetes or weight loss.
* Have had or are planning to have weight loss surgery.
* Have major health issues like severe kidney disease, untreated thyroid problems, or skin conditions where the glucose monitor would be placed.
* Have been part of another clinical trial recently.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Responder Rate | 6 Months
  Investigators will measure how many participants successfully reached their weight management goals by the end of 6 months. This 'Responder Rate' tells us the percentage of people in our study who effectively managed their weight using the methods we provided, whether it's through the Signos System or standard lifestyle education.
Average Total Body Weight Loss (TBWL%) | 6 Months
  Investigators will measure how much weight, on average, participants have lost after 6 months in the study. This will be calculated as a percentage of their initial weight. This measure helps us understand the effectiveness of the Signos System in helping participants reduce their body weight over a 6-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Kim, MD, Study Chair — Signos Inc
Locations (5):
- United States (5):
  - Helios Clinical Research (Phoenix), Phoenix, Arizona
  - Diablo Clinical Research, Walnut Creek, California
  - Segal Trials, North Miami, Florida
  - Helios Clinical Research, Houston, Texas
  - Seattle Clinical Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall H, Perelman D, Breschi A, Limcaoco P, Kellogg R, McLaughlin T, Snyder M. Glucotypes reveal new patterns of glucose dysregulation. PLoS Biol. 2018 Jul 24;16(7):e2005143. doi: 10.1371/journal.pbio.2005143. eCollection 2018 Jul. PMID 30040822
- [Background] Adams OP. The impact of brief high-intensity exercise on blood glucose levels. Diabetes Metab Syndr Obes. 2013;6:113-22. doi: 10.2147/DMSO.S29222. Epub 2013 Feb 27. PMID 23467903
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Baron AD. Impaired glucose tolerance as a disease. Am J Cardiol. 2001 Sep 20;88(6A):16H-9H. doi: 10.1016/s0002-9149(01)01832-x. PMID 11576521
- [Background] Brown A, McArdle P, Taplin J, Unwin D, Unwin J, Deakin T, Wheatley S, Murdoch C, Malhotra A, Mellor D. Dietary strategies for remission of type 2 diabetes: A narrative review. J Hum Nutr Diet. 2022 Feb;35(1):165-178. doi: 10.1111/jhn.12938. Epub 2021 Sep 1. PMID 34323335
- [Background] Chin SO, Keum C, Woo J, Park J, Choi HJ, Woo JT, Rhee SY. Successful weight reduction and maintenance by using a smartphone application in those with overweight and obesity. Sci Rep. 2016 Nov 7;6:34563. doi: 10.1038/srep34563. PMID 27819345
- [Background] Ebbeling CB, Knapp A, Johnson A, Wong JMW, Greco KF, Ma C, Mora S, Ludwig DS. Effects of a low-carbohydrate diet on insulin-resistant dyslipoproteinemia-a randomized controlled feeding trial. Am J Clin Nutr. 2022 Jan 11;115(1):154-162. doi: 10.1093/ajcn/nqab287. PMID 34582545
- [Background] Ehrhardt N, Al Zaghal E. Behavior Modification in Prediabetes and Diabetes: Potential Use of Real-Time Continuous Glucose Monitoring. J Diabetes Sci Technol. 2019 Mar;13(2):271-275. doi: 10.1177/1932296818790994. Epub 2018 Aug 1. PMID 30066574
- [Background] The Lancet Diabetes Endocrinology. Metabolic health: a priority for the post-pandemic era. Lancet Diabetes Endocrinol. 2021 Apr;9(4):189. doi: 10.1016/S2213-8587(21)00058-9. Epub 2021 Mar 4. No abstract available. PMID 33676599
- [Background] Galderisi A, Giannini C, Weiss R, Kim G, Shabanova V, Santoro N, Pierpont B, Savoye M, Caprio S. Trajectories of changes in glucose tolerance in a multiethnic cohort of obese youths: an observational prospective analysis. Lancet Child Adolesc Health. 2018 Oct;2(10):726-735. doi: 10.1016/S2352-4642(18)30235-9. Epub 2018 Aug 24. PMID 30236381
- [Background] Gonzalez-Rodriguez M, Pazos-Couselo M, Garcia-Lopez JM, Rodriguez-Segade S, Rodriguez-Garcia J, Tunez-Bastida C, Gude F. Postprandial glycemic response in a non-diabetic adult population: the effect of nutrients is different between men and women. Nutr Metab (Lond). 2019 Jul 17;16:46. doi: 10.1186/s12986-019-0368-1. eCollection 2019. PMID 31346341
- [Background] Guyenet SJ, Schwartz MW. Clinical review: Regulation of food intake, energy balance, and body fat mass: implications for the pathogenesis and treatment of obesity. J Clin Endocrinol Metab. 2012 Mar;97(3):745-55. doi: 10.1210/jc.2011-2525. Epub 2012 Jan 11. PMID 22238401
- [Background] Hamley S, Kloosterman D, Duthie T, Dalla Man C, Visentin R, Mason SA, Ang T, Selathurai A, Kaur G, Morales-Scholz MG, Howlett KF, Kowalski GM, Shaw CS, Bruce CR. Mechanisms of hyperinsulinaemia in apparently healthy non-obese young adults: role of insulin secretion, clearance and action and associations with plasma amino acids. Diabetologia. 2019 Dec;62(12):2310-2324. doi: 10.1007/s00125-019-04990-y. Epub 2019 Sep 6. PMID 31489455
- [Background] Hyde PN, Sapper TN, Crabtree CD, LaFountain RA, Bowling ML, Buga A, Fell B, McSwiney FT, Dickerson RM, Miller VJ, Scandling D, Simonetti OP, Phinney SD, Kraemer WJ, King SA, Krauss RM, Volek JS. Dietary carbohydrate restriction improves metabolic syndrome independent of weight loss. JCI Insight. 2019 Jun 20;4(12):e128308. doi: 10.1172/jci.insight.128308. eCollection 2019 Jun 20. PMID 31217353